CLINICAL TRIAL: NCT07144462
Title: A Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of NEUK203-215 Injection in Adult Chinese Patients With Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Neukio Biotherapeutics (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025SL066
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): NEUK203-215 Injection+Drug:Fludarabine+Drug:Cyclophosphamide
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide (C); Genetic: NEUK203-215 Injection

INTERVENTIONS:
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide (C) — Specified dose on specified days
Genetic: NEUK203-215 Injection — Specified dose on specified days

SUMMARY:
The purpose of this study is to determine the safety, tolerability and preliminary efficacy of NEUK203-215 , a healthy donor (HD) allogeneic CD19/BCMA-targeted CAR-NK cell product, in participants with severe, refractory autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* 1) Has provided signed informed consent; 2) Is aged 18-65 years ; 3)Adequate functional reserve of vital organs 4) Has a confirmed diagnosis of systemic lupus erythematosus, diffuse systemic sclerosis, inflammatory myopathy, or autoimmune bullous dermatosis.

Exclusion Criteria:

* 1) Requires dialysis treatment. 2) History of severe drug hypersensitivity. 3) Active infection requiring systemic therapy or suspected uncontrolled infection.

  4) Within 6 months before screening, any of the following cardiovascular events: New York Heart Association (NYHA) Class III or IV heart failure, myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmia, any ventricular arrhythmia, or other clinically significant cardiac disease.

  5) Malignancy within the past 5 years. 6) Clinically significant chronic or intermittent bleeding within 60 days before the screening visit.

  7) Prior solid-organ (e.g., heart, lung, kidney, liver) or hematopoietic stem-cell/bone-marrow transplantation.

  8) At screening: positive HBsAg and/or HBcAb with HBV DNA detectable or above the lower limit of quantitation; positive HCV antibody with HCV RNA detectable or above the lower limit of quantitation; positive HIV antibody; positive syphilis test (except biologic false-positive results).

  9) Major surgery within 4 weeks before screening. 10) Live or live-attenuated vaccine received within 4 weeks before screening. 11) Uncontrolled concurrent medical conditions. 12) Documented history of neurologic or psychiatric disorders. 13) Any other factor that, in the investigator's judgment, could require premature withdrawal from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-09-04 (Estimated); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 12 months post NEUK203-215 infusion
Existence/non existence of dose limiting toxicity (DLT) | Up to 12 months post NEUK203-215 infusion
serious adverse events (SAEs) | Up to 12 months post NEUK203-215 infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided